CLINICAL TRIAL: NCT07171970
Title: The Effectiveness and Safety of In Vitro Maturation With Fresh Embryo Transfer (The SAIGON Protocol) Versus In Vitro Fertilization With Frozen Embryo Transfer in Women With Polycystic Ovary Syndrome
Brief Title: IVM - Fresh ET (THE SAIGON PROTOCOL) Versus IVF - FET in PCOS Women
Acronym: SAIGON-PTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/25/DD-BVMD
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovary Syndrome (PCOS); In Vitro Maturation of Oocytes; Fresh Embryo Transfer
Keywords: in vitro maturation; The SAIGON protocol; fresh embryo transfer; GnRH-Antagonist; frozen embryo transfer
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVM-Fresh (No gonadotropin + Fresh embryo transfer) (Experimental): Endometrial preparation will be conducted using an artificial cycle protocol initiated on day 2-4 of the menstrual cycle (either spontaneous or induced). CAPA-IVM treatment will subsequently be performed, followed by oocyte fertilization and fresh embryo transfer.
  Interventions: Procedure: IVM-Fresh (No gonadotropin + Fresh embryo transfer)
- IVF-FET (GnRH-Antagonist - Agonist Trigger - Frozen embryo transfer) (Active Comparator): Ovarian stimulation will be performed using a GnRH-antagonist protocol starting on any day of the menstrual cycle. Embryos obtained from ICSI will be cryopreserved for later transfer.
  Interventions: Procedure: IVF-FET (GnRH-Antagonist - Agonist Trigger - Frozen embryo transfer)

INTERVENTIONS:
Procedure: IVM-Fresh (No gonadotropin + Fresh embryo transfer) — Patients randomized to this arm will receive estradiol valerate 8 mg/day. IVM will be performed after ≥10 days of estrogen and ET ≥8 mm. From the day of ICSI, they will continue estradiol and start vaginal progesterone 800 mg/day + dydrogesterone (20mg/day). A fresh embryo transfer will subsequently be performed.
  Arms: IVM-Fresh (No gonadotropin + Fresh embryo transfer)
Procedure: IVF-FET (GnRH-Antagonist - Agonist Trigger - Frozen embryo transfer) — Patients randomized into this group will receive FSH at a dose of 150 IU/day. Oocyte retrieval will be performed once the criteria for triggering are fulfilled, followed by embryo cryopreservation and frozen embryo transfer in the subsequent cycle. Endometrial preparation for frozen embryo transfer will be conducted using an exogenous steroids regimen. Patients will receive estradiol 8 mg/day starting from cycle days 2-3 for 10 days. When the endometrial thickness reaches ≥8 mm, luteal phase support will be initiated with vaginal progesterone 800 mg/day plus dydrogesterone 20 mg/day.
  Arms: IVF-FET (GnRH-Antagonist - Agonist Trigger - Frozen embryo transfer)

SUMMARY:
Assisted Reproductive Technologies (ART) aim to increase success rates while minimizing patient risks. For women with high AFC or PCOS, conventional IVF carries a high risk of OHSS (Ho et al., 2019). A modern IVF strategy to prevent this uses a GnRH agonist trigger, requiring a "freeze-all" and subsequent FET (Wong et al., 2017). This reduces OHSS risk but can increase time to pregnancy (Vuong et al., 2021) and treatment burden.

IVM is a patient-friendly alternative that eliminates OHSS risk by avoiding high-dose gonadotropins. A 2020 trial by Vuong et al. compared CAPA-IVM-FET to conventional IVF-FET in women with high AFC. IVM yielded a comparable live birth rate (35.2%) versus IVF (43.2%), with a 0% OHSS rate in IVM compared to 0.7% in IVF (Vuong et al., 2020).

The optimal transfer method (fresh or frozen) in IVM cycles is debated. A 2021 pilot RCT by Vuong et al. found a freeze-only strategy after CAPA-IVM led to a significantly higher live birth rate (60%) than a fresh transfer (20%) (Vuong et al., 2021), but increased time to pregnancy (194 vs. 150 days) (Vuong et al., 2021). A refined CAPA-IVM protocol, which uses no gonadotropins, allowed for fresh embryo transfer in the same cycle, resulting in a numerically higher ongoing pregnancy rate (43.3% vs. 33.3%) than FET (Vuong et al., 2025).

This raises an important question: how does a simplified IVM strategy with fresh transfer compare to the established "safety-net" IVF strategy with FET? These two approaches represent opposing clinical philosophies. No large-scale study has yet compared them in women with PCOS. Therefore, this study is designed to compare the SAIGON protocol (gonadotropin-free CAPA-IVM with fresh ET) against a standard GnRH-antagonist IVF protocol with agonist trigger and subsequent FET.

DETAILED DESCRIPTION:
1. Screening for eligibility and randomization: Women who are potentially eligible are provided with information about the trial. Screening is done on the day of the first visit, and patients are given informed consent form to sign before enrollment. Participants are then randomly assigned (1:1) to either the CAPA-IVM or IVF-FET group.
2. After randomisation 2.1. IVM-FRESH (The SAIGON Protocol):

   * Treatment begins on day 2-4 of the menstrual cycle.
   * Endometrial preparation uses oral estradiol valerate (Progynova®; Delpharm Lille SAS, France) 8mg/day for at least 10 days.
   * Immature oocyte retrieval is performed when the endometrial thickness is ≥ 8 mm.
   * Mature oocytes are fertilized via ICSI.
   * Luteal phase support is provided with vaginal progesterone (800 mg/day) + dydrogesterone (20mg/day) starting on the day of ICSI.
   * A fresh embryo transfer is performed three or five days after progesterone administration, depending on the embryo stage.

   2.2. IVF-FET (Frozen Transfer Protocol):
   * This protocol uses a random start approach, beginning on the day of the patient's first visit.
   * Ovarian stimulation is done using a GnRH antagonist protocol with a starting dose of 150 IU/day of rFSH.
   * A GnRH agonist trigger is administered when at least two leading follicles reach ≥ 17 mm in diameter.
   * Insemination is performed using ICSI for matured oocytes.
   * The endometrium is prepared for frozen embryo transfer using oral oestradiol valerate (8mg/day) and vaginal progesterone (800 mg/day) + dydrogesterone (20mg/day) when endometrial thickness is ≥ 8 mm.
   * Surviving embryos are thawed and transferred two hours after thawing under ultrasound guidance.
3. Pregnancy and outcomes:

   * A pregnancy test is performed 10-14 days after embryo transfer. A positive result is a serum hCG level of ≥ 25 mIU/mL.
   * Both groups continue hormone supplementation if the pregnancy test is positive.
   * The primary outcome of the study is the live birth rate after one embryo transfer. Secondary outcomes include cumulative ongoing pregnancy, time to ongoing pregnancy, clinical pregnancy rate, miscarriage, and other treatment and pregnancy complications.
   * Obstetric and neonatal outcomes: All data relating to the delivery process and neonatal care will be recorded by the data management system of IVFMD.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 - 42 years old.
* Diagnosed with PCOS, followed Rotterdam 2003 criteria (Group TREP consensus workshop, 2004)
* Had fewer than three previous failed frozen embryo transfer (FET) cycles
* Transferred no more than two cleavage embryos or one good-quality blastocyst or no more than two poor-quality blastocysts.
* Agreeing to participate in the study

Exclusion Criteria:

* Having allergy and contraindications for exogenous hormone administration (e.g., breast cancer, thromboembolic disease)
* Cycles with preimplantation genetic testing indication
* Oocyte donation cycles
* Having untreated uterine or adnexal abnormalities (e.g., intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus, large leiomyoma ≥5 cm in diameter; adenomyosis, endometrial polyp, hydrosalpinx).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Live birth rates after the one embryo transfer | At 24 weeks of gestation
  Live birth was defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. Live births refer to the individual newborn; for example, a twin delivery represents two live births.

SECONDARY OUTCOMES:
Cumulative ongoing pregnancy | After 12 months of follow-up after randomisation
  Cumulative ongoing pregnancy defined as the occurrence of at least one ongoing pregnancy within 12 months of follow-up after randomisation. An ongoing pregnancy is counted as 1 for each participant who achieves at least one such pregnancy within this time frame, regardless of the number of embryo transfers or pregnancies achieved. Participants who do not return for embryo transfer within the 12-month period are considered censored
Time to ongoing pregnancy | Up to 10 weeks after embryo placement
  Time to ongoing pregnancy defined as the interval between randomization and the achievement of an ongoing pregnancy.
Positive pregnancy test rate | 10-14 days after embryo transfer
  Positive pregnancy test rate defined as serum human chorionic gonadotropin level ≥ 25 mIU/mL.
Clinical pregnancy rate | 6 weeks after embryo transfer
  A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy.
Ongoing pregnancy rate | 12 weeks after embryo transfer
  A pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with a discernible heartbeat at 12 weeks gestation or beyond
Implantation rate | 3 weeks after embryo transfer
  The number of gestational sacs observed divided by the number of embryos transferred (usually expressed as a percentage)
Ectopic pregnancy rate | 2 - 4 weeks after embryo transfer
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Miscarriage rate | 2-22 weeks after embryo transfer
  Spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus.
Multiple gestations rate | 5 weeks after embryo transfer
  A pregnancy with more than one embryo or fetus
Multiple birth rate | At 22 weeks' gestation
  The complete expulsion or extraction from a woman of more than one fetus, after 22 completed weeks of gestational age, irrespective of whether it is a live birth or stillbirth. Births refer to the individual newborn; for example, a twin delivery represents two births.
Mode of delivery | At delivery
  Vaginal delivery, Assisted vaginal delivery, C-section
Birth weight | At delivery
  Weight of the newborn measured right after delivery
Gestational age at birth | At delivery
  Calculated by gestational age of all live births
Ovarian hyperstimulation syndrome | Up to 1 week after the oocyte retrieval in the IVF arm
  Ovarian hyperstimulation syndrome (OHSS) is a potentially lethal iatrogenic complication of the early luteal phase or/and early pregnancy after ovulation induction or ovarian stimulation. OHSS was evaluated if symptoms were reported by the patient.
IVM oocyte retrieval cancellation | After 21 day of endometrial preparation
  Record the reason for canceling in IVM arm
Embryo transfer cancellation | After 21 days of endometrial preparation
  Record the reason for canceling.
Preterm birth | At delivery
  Defined as delivery at <28, <32, <37 completed weeks. A birth that takes place after 22 weeks and before 37 completed weeks of gestational age.
Gestational diabetes mellitus | At 24-28 weeks of gestation
  A 75-g OGTT, with plasma glucose measurement when the patient is fasting and at 1 and 2 h, at 24-28 weeks of gestation in women not previously diagnosed with diabetes.
Hypertensive disorders of pregnancy | After 20 weeks of gestation
  Pregnancy-induced hypertension, pre-eclampsia (early and late), eclampsia, and HELLP syndrome
Stillbirth | At delivery after 28 weeks of gestation
  The death of a fetus before the complete expulsion or extraction from its mother after 28 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles. It includes deaths occurring during labor.
Very low birth weight | At delivery
  Birth weight less than 1.500 g.
Low birth weight | At delivery
  Birth weight less than 2.500 g
High birth weight | At delivery
  Implies growth beyond an absolute birth weight of 4.000 g, regardless of the gestational age
Very high birth weight | At delivery
  Birth weight over 4.500 g.
Major congenital abnormalities | During pregnancy and 12 months after delivery
  Structural, functional, and genetic anomalies that occur during pregnancy, and are identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or life-threatening, or cause death. Any congenital anomaly will be included as follows definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
Postpartum hemorrhage | Up to one month after the delivery
  Defined as a blood loss of ≥ 1000 mL, or blood loss accompanied by signs or symptoms of hypovolemia, within 24 hours after birth (including intrapartum blood loss), regardless of the mode of delivery.
NICU admission | Up to one month after the delivery
  The admission of the newborn to the NICU
Neonatal mortality | Up to one month after the delivery
  Death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between 8 and 28 days after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- IVFMD - My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No